CLINICAL TRIAL: NCT06843720
Title: Expanding Access to Cervical Cancer Screening Through Primary HR-HPV Testing and Self-sampling: a Multicomponent Intervention for Safety Net Health Systems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024-0361; NCI-2025-01326 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: HR-HPV Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Participants participate in an interview or a focus group discussion and provide opinions about self-collection and/or education and training materials for participants and providers.
  Partipants participation in this study may be limited to a single interview or focus group discussion. Some stakeholders will be asked to participate in additional interviews and/or focus groups.
  Interventions: Behavioral: HR-HPV Testing

INTERVENTIONS:
Behavioral: HR-HPV Testing — Given by Interview and focus groups

SUMMARY:
To learn about the attitudes toward implementing self-collection among healthcare providers and staff, participants, and other stakeholders; and to inform the development of patient education and provider training materials to aid in the implementation of self-collection in clinical settings.

DETAILED DESCRIPTION:
The overarching goal of the implementation program is to increase cervical cancer screening, early detection, and linkage to treatment in underserved populations that receive care in safety net health systems. Specific goals are:

1. To increase up-to-date cervical cancer screening coverage by 10%;
2. To increase clinical encounters used for opportunistic cervical cancer screening using primary HR-HPV testing by 5% annually;
3. To increase awareness and readiness for implementing primary HR-HPV testing with self-sampling in routine care among clinics in the ECHO Network;
4. All patrticipants with abnormal screening results will be navigated to and receive diagnostic testing.

The overarching goal of program evaluation (i.e., research component of this protocol) is to evaluate the progress and achievement of program goals and to evaluate effectiveness and implementation outcomes:

Primary objective 1: Evaluate the effectiveness of primary HPV testing and self-collection to increase participation in cervical cancer screening among underscreened health system participants.

Primary objective 2: Evaluate implementation outcomes of the program across health systems and clinics and explore mechanisms underlying outcomes, guided by the Consolidated Framework for Implementation Research (CFIR)41,42 and RE-AIM (reach, effectiveness, adoption, implementation, maintenance)43.

Secondary Objectives Secondary objective 1: Compare the proportion of clinical encounters used for opportunistic cervical cancer screening across clinics.

Secondary objective 2: Evaluate proportion of participants receiving clinical follow-up after a positive HR-HPV test.

Secondary objective 3: Describe the prevalence of cervical cancer and pre-cancer among participants who self-collected and tested positive for HR-HPV.

Secondary objective 4: Compare the effectiveness of clinic-based primary HPV testing with self-collection with and without preceding telephone-based patient education by a participant navigator.

ELIGIBILITY:
Inclusion Criteria:

Populations involved in the research are: 1) stakeholder advisory board members; 2) Participants eligible for cervical cancer screening participating in the cluster randomized stepped-wedge trial; 3) Patients and community members participating in formative research activities; 4) Investigators, clinic staff, and other health system stakeholders from partnering health systems; 5) Project ECHO Participants (providers, clinic staff, and other health system stakeholders from partner and non-partner institutions).

The eligibility criteria for each are:

Participants eligible for cervical cancer screening:

* Currently a resident in the state of Texas
* Attend for care at a partner clinic enrolled in the study
* Women and persons with a cervix
* Age 25-65
* Due or past due for cervical cancer screening

Participants and community members participating in formative research activities:

* Purposively identified as a stakeholder for formative research by research staff Investigators, clinic staff, and other health system stakeholders from partnering health systems:
* Employed at least part-time by a partnering health system
* Age 18+

Project ECHO Participants:

* Participate in at least one Project ECHO session
* Age 18+

Exclusion Criteria:

Participants eligible for cervical cancer screening:

* Report being currently pregnant
* History of total hysterectomy
* History of cervical cancer

Other study populations:

• Unable to communicate in English or Spanish

Vulnerable Populations Participants/samples belonging to vulnerable populations (children, pregnant women, cognitively impaired adults, or prisoners) will be prohibited from participation.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 7100 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs). Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 4.03 | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org